CLINICAL TRIAL: NCT03936660
Title: COOrdinating CaRDIology CliNics RAndomized Trial of Interventions to Improve OutcomEs (COORDINATE) - Diabetes
Brief Title: A 12 Month Site Randomized Trial in Adults With Type 2 Diabetes Mellitus and History of Cardiovascular Disease
Acronym: COORDINATE
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Duke University (Other)
Collaborators: Boehringer Ingelheim (Industry); Eli Lilly and Company (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Health Services Research
Other Study IDs: Pro00101556
Record Dates: First submitted 2019-05-01; First posted 2019-05-03 (Actual); Results first posted 2024-11-21 (Actual); Last update posted 2024-11-21 (Actual); Status verified 2024-04

CONDITIONS: Diabetes Mellitus, Type 2; Cardiovascular Diseases
Keywords: COORDINATE-DIABETES; COORDINATE; T2DM; Diabetes Mellitus, Type 2; Cardiovascular Disease; Prevention
MeSH Terms: conditions — Diabetes Mellitus, Type 2; Cardiovascular Diseases | interventions — Methods

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Control (No Intervention): Clinics provided with existing clinical care guidelines.
- Intervention (Active Comparator): Clinics provided with existing clinical care guidelines as well as a multifaceted educational intervention to support development of an integrated, multi-disciplinary care pathway for patients with T2DM and CVD.
  Interventions: Other: Intense Education Intervention

INTERVENTIONS:
Other: Intense Education Intervention — Clinics provided with existing clinical care guidelines as well as a multifaceted educational intervention to support development of an integrated, multi-disciplinary care pathway for patients with T2DM and CVD.
  Other Names: Intervention
  Arms: Intervention

SUMMARY:
COORDINATE-Diabetes is a cluster-randomized clinical trial to test the effectiveness of an innovative, clinic-level educational intervention to improve the management of patients with type 2 diabetes mellitus and cardiovascular disease.

DETAILED DESCRIPTION:
Patients with Type 2 diabetes mellitus and a history of cardiovascular disease will be enrolled in this study. The study will randomize a minimum of 42 US cardiology clinics to an intervention arm vs. control arm. The clinic-level multi-faceted educational intervention will include strategies to develop cardiology and endocrinology partnerships and guideline-recommended care pathways with measurement and feedback to improve the care of patients with type 2 diabetes mellitus and cardiovascular disease.

Patients must be enrolled during a routine visit in a cardiology clinic, and the clinic must have at least 3 physicians and/or APPs on staff with independent patient populations.

ELIGIBILITY:
Inclusion Criteria:

* Age ≥ 18 years old
* Diagnosis of Type 2 diabetes mellitus (T2DM)
* History of at least one of the following conditions:

  1. Coronary artery disease (defined as prior MI, coronary revascularization (CABG or PCI), and/or obstructive CAD (≥50%) as documented by angiography or CTA)
  2. Stroke and/or carotid artery stenosis (≥50%)
  3. Peripheral Arterial disease (defined as claudication with ABI<0.9, prior peripheral revascularization, and/or amputation due to circulatory insufficiency)
* Ability to communicate with site staff and understand and provide written informed consent and proof of Health Insurance Portability and Accountability Act (HIPAA) authorization

Exclusion Criteria:

* Determined to be highly unlikely to survive and/or to continue follow-up in that clinic for at least 1 year, as identified by site investigator
* GFR<30 mL/min/1.73m2
* Already on all guideline-recommended therapies for T2DM and CVD
* Absolute contraindication to any of the guideline recommended therapies for T2DM and CVD

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 1049 (Actual)
Dates: Start 2019-07-25 (Actual); Primary Completion 2022-12-30 (Actual); Study Completion 2022-12-30 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Christopher Granger, MD, Principal Investigator — Duke Clinical Research Institute
Locations (44):
- United States (44):
  - Grandview Health/Alabama Cardiovascular Group, Birmingham, Alabama
  - USA Cardiology, Mobile, Alabama
  - Alaska Heart and Vascular Institute, Anchorage, Alaska
  - Dignity Health/DHMG Specialty Medicine, Phoenix, Arizona
  - Stanford University, Stanford, California
  - Blue Coast Cardiology, Vista, California
  - Aurora Denver Cardiology, Denver, Colorado
  - Bridgeport Hospital, Bridgeport, Connecticut
  - Orlando Heart and Vascular Institute, Altamonte Springs, Florida
  - Riverside Medical Center/Synergy Healthcare, Bradenton, Florida
  - Lennar Foundation/Univ. of Miami, Coral Gables, Florida
  - Citrus Cardiology, Inverness, Florida
  - Baptist Health Research Institute, Jacksonville, Florida
  - Advanced Research for Health Improvement, LLC, Naples, Florida
  - Cardiovascular Inst. of Northwest Florida, Panama City, Florida
  - Bayfront Cardiovascular Associates, St. Petersburg, Florida
  - Interventional Cardiac Consultants, Trinity, Florida
  - Emory/Grady Memorial Hospital, Atlanta, Georgia
  - Advocate Heart Institute, Chicago, Illinois
  - Advanced Heart Care Group/Medicoricium LLC, Fairview Heights, Illinois
  - Specialty Physicians of Illinois, Olympia Fields, Illinois
  - UnityPoint Health Cardiovascular Services, Peoria, Illinois
  - Prairie Cardiovascular Consultants, Springfield, Illinois
  - Iowa Heart Center, Des Moines, Iowa
  - Heart Clinic of Louisiana, Marrero, Louisiana
  - The Johns Hopkins University, Baltimore, Maryland
  - Endeavor Medical Research, Alpena, Michigan
  - Cardiology Institute of Michigan, Flint, Michigan
  - Hannibal Regional Medical Group, Hannibal, Missouri
  - Advanced Heartcare LLC, Bridgewater, New Jersey
  - New Jersey Heart, Linden, New Jersey
  - Garden State Heart Care, Manalapan, New Jersey
  - Cardiovascular Associates of the Delaware Valley, Sewell, New Jersey
  - Northwell Health/Lenox Hill Hospital, Manhasset, New York
  - Kernodle Clinic, Burlington, North Carolina
  - Cone Health/LeBauer Brodie Ctr for Cardiovascular Rsch, Greensboro, North Carolina
  - Cape Fear Heart Associates, Wilmington, North Carolina
  - Cardiovascular Health Clinic, Oklahoma City, Oklahoma
  - Guthrie Medical Group, Sayre, Pennsylvania
  - Advanced Cardiology Associates, Greenwood, South Carolina
  - Black Hills Cardiovascular Research, Rapid City, South Dakota
  - Univ. of Texas Southwestern, Dallas, Texas
  - Lonestar Heart and Vascular, Tomball, Texas
  - ProHealth Care Heart and Vascular, Waukesha, Wisconsin

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Zinman B, Lachin JM, Inzucchi SE. Empagliflozin, Cardiovascular Outcomes, and Mortality in Type 2 Diabetes. N Engl J Med. 2016 Mar 17;374(11):1094. doi: 10.1056/NEJMc1600827. No abstract available. PMID 26981940
- [Background] Marso SP, Daniels GH, Brown-Frandsen K, Kristensen P, Mann JF, Nauck MA, Nissen SE, Pocock S, Poulter NR, Ravn LS, Steinberg WM, Stockner M, Zinman B, Bergenstal RM, Buse JB; LEADER Steering Committee; LEADER Trial Investigators. Liraglutide and Cardiovascular Outcomes in Type 2 Diabetes. N Engl J Med. 2016 Jul 28;375(4):311-22. doi: 10.1056/NEJMoa1603827. Epub 2016 Jun 13. PMID 27295427
- [Background] Sattar N, Petrie MC, Zinman B, Januzzi JL Jr. Novel Diabetes Drugs and the Cardiovascular Specialist. J Am Coll Cardiol. 2017 May 30;69(21):2646-2656. doi: 10.1016/j.jacc.2017.04.014. PMID 28545639
- [Background] Vinereanu D, Lopes RD, Bahit MC, Xavier D, Jiang J, Al-Khalidi HR, He W, Xian Y, Ciobanu AO, Kamath DY, Fox KA, Rao MP, Pokorney SD, Berwanger O, Tajer C, de Barros E Silva PGM, Roettig ML, Huo Y, Granger CB; IMPACT-AF investigators. A multifaceted intervention to improve treatment with oral anticoagulants in atrial fibrillation (IMPACT-AF): an international, cluster-randomised trial. Lancet. 2017 Oct 14;390(10104):1737-1746. doi: 10.1016/S0140-6736(17)32165-7. Epub 2017 Aug 28. PMID 28859942
- [Background] American Diabetes Association. 9. Pharmacologic Approaches to Glycemic Treatment: Standards of Medical Care in Diabetes-2019. Diabetes Care. 2019 Jan;42(Suppl 1):S90-S102. doi: 10.2337/dc19-S009. PMID 30559235
- [Background] American Diabetes Association. 10. Cardiovascular Disease and Risk Management: Standards of Medical Care in Diabetes-2019. Diabetes Care. 2019 Jan;42(Suppl 1):S103-S123. doi: 10.2337/dc19-S010. PMID 30559236
- [Derived] Tannu M, Kaltenbach L, Pagidipati NJ, McGuire DK, Aroda VR, Pop-Busui R, Kondamudi N, Al-Khalidi HR, Lopes RD, Cavender MA, Nelson AJ, Kirk J, Lingvay I, Magwire M, Richardson CR, Webb L, Leyva M, Pandey A, Washington A, Pak J, Gaynor T, Khan W, Weston P, Granger CB, Green J. Effects of an Intervention to Improve Evidence-Based Care for People With Diabetes and Cardiovascular Disease Across Sex, Race, and Ethnicity Subgroups: Insights From the COORDINATE-Diabetes Trial. Circulation. 2024 Jul 16;150(3):180-189. doi: 10.1161/CIRCULATIONAHA.124.068962. Epub 2024 Jun 27. PMID 38934111
- [Derived] Pagidipati NJ, Nelson AJ, Kaltenbach LA, Leyva M, McGuire DK, Pop-Busui R, Cavender MA, Aroda VR, Magwire ML, Richardson CR, Lingvay I, Kirk JK, Al-Khalidi HR, Webb L, Gaynor T, Pak J, Senyucel C, Lopes RD, Green JB, Granger CB; COORDINATE-Diabetes Site Investigators. Coordinated Care to Optimize Cardiovascular Preventive Therapies in Type 2 Diabetes: A Randomized Clinical Trial. JAMA. 2023 Apr 18;329(15):1261-1270. doi: 10.1001/jama.2023.2854. PMID 36877177

RESULTS

PARTICIPANT FLOW:
Units Other Than Participants: Sites
Groups:
- Intervention: Provided with existing clinical care guidelines as well as a multifaceted educational intervention to support development of an integrated, multi-disciplinary care pathway for patients with T2DM and CVD.
- Control: Provided with existing clinical care guidelines.
Period: Overall Study
Arm/Group | Intervention | Control
Started | 459; 25 Sites | 590; 24 Sites
Completed | 457; 20 Sites (25 sites randomized, of which, 5 sites dropped out prior to enrolling participants.) | 588; 23 Sites (24 sites randomized, of which, 1 site dropped out prior to enrolling participants.)
Not Completed | 2; 5 Sites | 2; 1 Sites
Not completed — Missing medication data at 6 and 12 months. | 2 | 2

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Intervention | Control | Total
Number analyzed (Participants) | 459 | 590 | 1049
Age, Continuous [Median (Inter-Quartile Range); unit: years] | 69 [63 to 76] | 71 [64 to 77] | 70 [63 to 76]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 144 | 194 | 338
  Male | 315 | 396 | 711
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 52 | 38 | 90
  Not Hispanic or Latino | 391 | 550 | 941
  Unknown or Not Reported | 16 | 2 | 18
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 1 | 6 | 7
  Asian | 17 | 10 | 27
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 79 | 93 | 172
  White | 324 | 477 | 801
  More than one race | 0 | 0 | 0
  Unknown or Not Reported | 38 | 4 | 42
Health Insurance [Count of Participants; unit: Participants]
  Medicare (alone or with other insurance) | 282 | 410 | 692
  Private only | 114 | 109 | 223
  Medicaid only | 34 | 31 | 65
  Other insurance only | 18 | 28 | 46
  No insurance | 11 | 12 | 23
Baseline Composite Medication Score [Count of Participants; unit: Participants] — Number of recommended medications being taken by the participant at baseline.
  Participants
    0 points (not taking any recommended medications) | 27 | 57 | 84
    1 point (taking one recommended medication) | 157 | 226 | 383
    2 points (taking two recommended medications) | 275 | 307 | 582

OUTCOME MEASURES:

1. Primary Outcome: Number of Participants Prescribed All 3 Groups of Recommended Evidence-based Medications
Description: Proportion of patients prescribed all three groups of guideline-recommended therapies for management for T2DM and CVD at last follow-up visit. Groups were defined as (1) high-intensity statins (40-80 mg/d atorvastatin or 20-40 mg/d rosuvastatin); (2) ACEIs or ARBs including angiotensin receptor-neprilysin inhibitors (ARNIs); and (3) SGLT2 inhibitors and/or GLP-1RAs with proven cardiovascular benefit (SGLT2 inhibitors: empagliflozin, dapagliflozin, or canagliflozin; GLP-1RAs: liraglutide, semaglutide, or dulaglutide), or metformin monotherapy with hemoglobin A1c < 7%.
Time Frame: Up to 12 Months
Population: All participants for whom medication data was available at 6 or 12 months.
Measure: Count of Participants; unit: Participants
Arm/Group | Intervention | Control
Number analyzed (Participants) | 457 | 588
Participants | 173 | 85

2. Secondary Outcome: Number of Participants on Guideline Recommended Therapies at Last Follow-up Visit.
Description: Number of participants prescribed each of the 3 recommended therapies at the last follow-up visit.
Time Frame: Up to 12 Months
Population: All participants for whom medication data was available at 6 or 12 months.
Measure: Count of Participants; unit: Participants
Arm/Group | Intervention | Control
Number analyzed (Participants) | 457 | 588
Participants
  Prescribed high-intensity statin | 323 | 334
  Prescribed ACEI or ARB | 372 | 402
  Prescribed SGLT-2i and/or GLP-1RA | 276 | 209
  Prescribed 2 or more groups of recommended medications (composite score >= 2) | 361 | 326
  Prescribed all 3 groups (without metformin monotherapy option) | 142 | 50

3. Secondary Outcome: Change in Average LDL-C From Baseline to Last Follow-up Visit.
Description: Average change in LDL-C values between baseline visit and last follow-up visit.
Time Frame: Baseline and last follow-up visit (up to 12 months)
Population: All participants for whom medication data was available at 6 or 12 months, and who had cholesterol data available at baseline and last follow-up.
Measure: Mean (Standard Error); unit: mg/dL
Arm/Group | Intervention | Control
Number analyzed (Participants) | 244 | 211
mg/dL
  Baseline | 72.93 (33.7) | 75.07 (30.66)
  Last follow-up visit | 68.79 (31.17) | 70.60 (32.96)

4. Secondary Outcome: Number of Participants With LDL-C < 70 mg/dL
Description: Change in number of participants with LDL-C < 70 mg/dL at baseline visit vs. last follow-up visit.
Time Frame: Baseline and last follow-up visit (up to 12 months)
Population: Participants with outcome data available at both baseline and last follow-up visit.
Measure: Number; unit: participants
Arm/Group | Intervention | Control
Number analyzed (Participants) | 244 | 213
participants
  Baseline | 131 | 111
  Last follow-up visit | 147 | 126

5. Secondary Outcome: Change in Average Blood Pressure From Baseline to Last Follow-up Visit.
Description: Change in systolic and diastolic blood pressure from baseline to last follow-up visit.
Time Frame: Baseline and last follow-up visit (up to 12 months)
Population: All participants for whom medication data was available at 6 or 12 months, who had systolic and diastolic blood pressure data at baseline and last follow-up visit.
Measure: Mean (Standard Error); unit: mmHg
Arm/Group | Intervention | Control
Number analyzed (Participants) | 377 | 486
mmHg
  Baseline systolic blood pressure | 131.40 (16.14) | 129.47 (16.48)
  Follow-up systolic blood pressure | 129.09 (17.36) | 130.35 (17.00)
  Baseline diastolic blood pressure | 74.04 (10.28) | 72.35 (10.90)
  Follow-up diastolic blood pressure | 72.44 (10.67) | 72.01 (11.28)

6. Secondary Outcome: Number of Participants With sBP < 130 mmHg
Description: Proportion of participants achieving sBP < 130 mmHg at baseline vs. last follow-up visit
Time Frame: Baseline and last follow-up visit (up to 12 months)
Population: Participants with outcome data available at both baseline and last follow-up visits
Measure: Number; unit: participants
Arm/Group | Intervention | Control
Number analyzed (Participants) | 378 | 492
participants
  Baseline | 185 | 243
  Last follow-up visit | 200 | 252

7. Secondary Outcome: Number of Participants With dBP < 180 mmHg
Description: Change in number of participants with dBP < 180 mmHg from baseline to last follow-up visit
Time Frame: Baseline and last follow-up visit (up to 12 months)
Population: Participants with outcome data available at both baseline and last follow-up visit
Measure: Number; unit: participants
Arm/Group | Intervention | Control
Number analyzed (Participants) | 378 | 498
participants
  Baseline | 271 | 348
  Last follow-up visit | 267 | 355

8. Secondary Outcome: Change in Average HbA1c From Baseline to Last Follow-up Visit.
Description: Change in hemoglobin A1c (HbA1c) between baseline and last follow-up visit.
Time Frame: Baseline and last follow-up visit (up to 12 months)
Population: All participants for whom medication data was available at 6 or 12 months, and who had HbA1c values available at baseline and last follow-up visit.
Measure: Mean (Standard Error); unit: HbA1c %
Arm/Group | Intervention | Control
Number analyzed (Participants) | 265 | 237
HbA1c %
  HbA1c at baseline | 7.64 (1.49) | 7.50 (1.40)
  HbA1c at last follow-up visit | 7.47 (1.67) | 7.49 (1.43)

9. Secondary Outcome: Number of Participants With HbA1c < 7%
Description: Change in number of participants with HbA1c < 7% from baseline to last follow-up visit.
Time Frame: Baseline and last follow-up visit (up to 12 months)
Population: Participants with outcome data available at both baseline and last follow-up visit
Measure: Number; unit: participants
Arm/Group | Intervention | Control
Number analyzed (Participants) | 265 | 239
participants
  Baseline | 181 | 169
  Last follow-up visit | 197 | 167

10. Secondary Outcome: Number of Participants Experiencing an Event Within 1 Year
Description: Number of participants experiencing an event within 12 months of enrollment. Also known as cumulative incidence of events.
Time Frame: Up to 12 Months
Population: All participants for whom medication data was available at 6 or 12 months.
Measure: Number; unit: participants
Arm/Group | Intervention | Control
Number analyzed (Participants) | 457 | 588
participants
  Composite (all-cause mortality, MI, stroke, urgent revascularization, decompensated HF) | 23 | 40
  All-cause mortality | 6 | 16
  Hospitalization for myocardial infarction (MI) | 3 | 3
  Hospitalization for stroke | 1 | 3
  Hospitalization for urgent revascularization | 8 | 7
  Hospitalization for decompensated heart failure (HF) | 8 | 18

ADVERSE EVENTS:
Time Frame: Up to 12 months.
Description: Per protocol, each site reported adverse events to Boehringer-Ingelheim (BI)'s pharmacovigilance team. Not all end point data were reported as adverse events.
Arm/Group | Intervention | Control
All-Cause Mortality (participants affected / at risk) | 6/459 | 16/590
Serious Adverse Events (participants affected / at risk) | 3/459 | 0/590
Other Adverse Events (participants affected / at risk) | 4/459 | 1/590
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Intervention (N=459) | Control (N=590)
Urinary tract infection (Infections and infestations) | 1 (1) | 0 (0)
Hyperglycaemic hyperosmolar nonketotic syndrome (Metabolism and nutrition disorders) | 1 (1) | 0 (0)
Acute kidney injury (Infections and infestations) | 1 (1) | 0 (0)
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Intervention (N=459) | Control (N=590)
Urinary tract infection (Infections and infestations) | 1 (1) | 0 (0)
Inflammation (General disorders) | 0 (0) | 1 (1)
Mental status changes (Infections and infestations) | 1 (1) | 0 (0)
Hypoglycemia (Infections and infestations) | 1 (1) | 0 (0)
Fungal infection (Infections and infestations) | 1 (1) | 0 (0)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (2):
  • Study Protocol (2021-10-25): https://cdn.clinicaltrials.gov/large-docs/60/NCT03936660/Prot_000.pdf
  • Statistical Analysis Plan (2022-06-16): https://cdn.clinicaltrials.gov/large-docs/60/NCT03936660/SAP_001.pdf